CLINICAL TRIAL: NCT06725043
Title: Ultrasound Acupuncture for Oxaliplatin-induced Peripheral Neuropathy in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Ali Mahmoud Ibrahim Badr Al-din, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ultrasound Acupuncture for OIP
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Patients and Their Partners; Oxaliplatin-induced Peripheral Neuropathy
Keywords: oxaliplatin; peripheral neuropathy; ultrasound acupuncture
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Therapeutic ultrasound (1 MHz) Pulsed mode at bilateral acupuncture points of PC6, PC7, BL60 andKI1
  Interventions: Device: Therapeutic ultrasound; Other: Traditional physical therapy program
- Experime (Placebo Comparator): Placebo Therapeutic ultrasound at bilateral acupuncture points of PC6, PC7, BL60, and KI1
  Interventions: Device: Placebo therapeutic ultrasound; Other: Traditional physical therapy program

INTERVENTIONS:
Device: Therapeutic ultrasound — Pulsed therapeutic ultrasound (1 MHz , 50% duty cycle and intensity gradually increased till the patient felt a deqi sensation).Each point was stimulated by ultrasound for 5 minutes at bilateral acupuncture points of PC6, PC7, BL60 and KI1(3 times / week for 4 weeks).
  Arms: Active
Device: Placebo therapeutic ultrasound — patients were received placebo therapeutic ultrasound at bilateral acupuncture points of PC6, PC7, BL60, and KI.
  Arms: Experime
Other: Traditional physical therapy program — Strengthing exercise, balance training, stretching exercises and home exercise program and education

SUMMARY:
The current study was conducted to examine the effect of ultrasound acupuncture for oxaliplatin-induced peripheral neuropathy in colorectal cancer patients.

DETAILED DESCRIPTION:
Oxaliplatin is platinum-based chemotherapy most usually used for the treatment of metastatic colorectal cancer, this drug can produce a cumulative and dose-limiting distal sensory neuropathy affecting the majority of oxaliplatin-treated patients. Despite intense investigation at the preclinical and clinical levels, no treatment can be suggested for the prevention of OIPN. Since acupuncture has proven effective in alleviating the severity of peripheral nerve neuropathy, as has ultrasound.

This systematic review was conducted to test the ability of ultrasound acupuncture in decreasing neuropathy-related symptoms induced by oxaliplatin-based chemotherapies in colorectal cancer patients

ELIGIBILITY:
Inclusion Criteria:

-

The subject selection was according to the following criteria:

* Adults their ages ranged from 20 to 70 years old.
* Receiving or have received chemotherapy treatment for colon or rectal cancer.
* Chemotherapy regimen included the agent oxaliplatin.
* Patients diagnosed with neuropathy by the oncologist.
* Both sexes.
* No neuropathy prior to oxaliplatin treatment.
* No documented or observable psychiatric or neurological disorders that would interfere with study participation (eg, dementia or psychosis)
* Stage II, III and IV colon or rectal cancer.
* Hands and Feets were the most affected by CIPN.
* The first dose of oxaliplatin was from 4 months or more.

Exclusion Criteria:

* The potential participants were excluded in the following conditions:

  * Another malignancy
  * Patients with severe or unstable cardiorespiratory or musculoskeletal diseases that may influence the accuracy of quantitative sensory testing results.
  * Participants who cannot remain on the same medications throughout the study period with minor dose adjustments allowed.
  * Contraindications to therapeutic ultrasound including active cancer in region of hands or feet, presence of deep vein thrombosis, complete numbness in hands or feet (representing severe CIPN), metal or plastic implantation
  * Peripheral vascular disease in hands or feet.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Pain level assessment | 2.5 months
  In comfortable siting position we asked them to give each item from the 10-items score from 0 to 10 according to the intensity of the symptom, 0 means that the symptom is absent and 10 means maximum intensity. Sum of scores is 100, a higher score is associated with increased pain
Assessment of pain pressure threshold | 2.5 months
  Pain pressure threshold at hand and foot was measured by using a digital pressure algometer with a probe of 1 cm2 .PPT at feets was measured on the plantar foot surface over the second metatarsal. PPT at hands was measured on thenar eminence of the hand

SECONDARY OUTCOMES:
National Cancer Institute Common Toxicity Criteria | 2.5 months
  NCI CTC are set of medical terms very useful for the classification of adverse events related to cytotoxic drugs. These terms are not international codes for reporting adverse events to the Health Authorities. They are very frequently used in handling adverse events from oncology trials

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Suez Canal University, Ismailia, Ismalia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol